CLINICAL TRIAL: NCT03380455
Title: A Single-center, Open-label Study to Investigate the Effect of Cimetidine on the Pharmacokinetics of Lucerastat in Healthy Male Subjects
Brief Title: Effect of Cimetidine on the Pharmacokinetics of Lucerastat in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-069-105
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — migalastat; Cimetidine

STUDY DESIGN:
Intervention Model Description: Fixed sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment period A & B (Experimental): Treatment period A: Subjects receive a single oral dose of 500 mg lucerastat on Day 1 under fasted conditions.
  Treatment period B: From Day 3 to Day 9, subjects receive a b.i.d. (every 12 h) oral dose of 800 mg cimetidine under fasted conditions (Treatment period B1; from Day 3 to Day 5). On Day 6, subjects receive a single oral dose of 500 mg lucerastat concomitantly with the morning dose of 800 mg cimetidine under fasted conditions (Treatment period B2; from Day 6 to Day 10).
  Interventions: Drug: Lucerastat; Drug: Cimetidine

INTERVENTIONS:
Drug: Lucerastat — Single oral dose of 500 mg lucerastat under fasted conditions
Drug: Cimetidine — Twice daily oral dose of 800 mg cimetidine under fasted conditions

SUMMARY:
A study in healthy male subjects to investigate whether repeated administrations of cimetidine (a medication which decreases the amount of acid in the stomach) can affect the fate in the body (amount and time of presence in the blood) of lucerastat. Safety of the concomitant administration of the two treatments will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Body mass index from 18.0 to 30.0 kg/m2 (inclusive) at Screening.
* Normal renal function confirmed by creatinine clearance ≥ 80 mL/min using Cockroft-Gault formula at Screening.

Exclusion Criteria:

* Known hypersensitivity to cimetidine, lucerastat, or drugs of the same class, or any of their excipients.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study treatment(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Cmax of lucerastat | Up to 48 h after lucerastat administration on Day 1 (i.e., up to Day 3) and from pre-dose up to 96 h after lucerastat administration on Day 6 (i.e., up to Day 10); in total for up to 7 days
  Plasma PK parameter of lucerastat after single-dose oral administration of lucerastat alone and in combination with cimetidine
Tmax of lucerastat | Up to 48 h after lucerastat administration on Day 1 (i.e., up to Day 3) and from pre-dose up to 96 h after lucerastat administration on Day 6 (i.e., up to Day 10); in total for up to 7 days
  Plasma PK parameter of lucerastat after single-dose oral administration of lucerastat alone and in combination with cimetidine
AUC(0-t) of lucerastat | Up to 48 h after lucerastat administration on Day 1 (i.e., up to Day 3) and from pre-dose up to 96 h after lucerastat administration on Day 6 (i.e., up to Day 10); in total for up to 7 days
  Plasma PK parameter of lucerastat after single-dose oral administration of lucerastat alone and in combination with cimetidine
AUC(0-inf) of lucerastat | Up to 48 h after lucerastat administration on Day 1 (i.e., up to Day 3) and from pre-dose up to 96 h after lucerastat administration on Day 6 (i.e., up to Day 10); in total for up to 7 days
  Plasma PK parameter of lucerastat after single-dose oral administration of lucerastat alone and in combination with cimetidine
AUC(0-48) of lucerastat | Up to 48 h after lucerastat administration on Day 1 (i.e., up to Day 3) and from pre-dose up to 96 h after lucerastat administration on Day 6 (i.e., up to Day 10); in total for up to 7 days
  Plasma PK parameter of lucerastat after single-dose oral administration of lucerastat alone and in combination with cimetidine
T1/2 of lucerastat | Up to 48 h after lucerastat administration on Day 1 (i.e., up to Day 3) and from pre-dose up to 96 h after lucerastat administration on Day 6 (i.e., up to Day 10); in total for up to 7 days
  Plasma PK parameter of lucerastat after single-dose oral administration of lucerastat alone and in combination with cimetidine

SECONDARY OUTCOMES:
Number of treatment-emergent AEs | From Day 1 to End-of-Study (for up to 13 days)
Number of treatment-emergent SAEs | From Screening to safety follow-up, i.e., 32 days after End-of-Study (for up to 63 days)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Boof, PhD, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

REFERENCES:
- [Derived] Boof ML, Halabi A, Ufer M, Dingemanse J. Impact of the organic cation transporter 2 inhibitor cimetidine on the single-dose pharmacokinetics of the glucosylceramide synthase inhibitor lucerastat in healthy subjects. Eur J Clin Pharmacol. 2020 Mar;76(3):431-437. doi: 10.1007/s00228-019-02808-9. Epub 2019 Dec 13. PMID 31836927